CLINICAL TRIAL: NCT06674434
Title: Comparative Effects of Sustained Stretch and Mobilization With Movement on Pain, Range of Motion, Muscle Strength and Functional Disability in Patient With Tennis Elbow.
Brief Title: Comparative Effects of Sustained Stretch and Mobilization With Movement in Patient With Tennis Elbow
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ RCR & AHS/24/0133
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
Keywords: Lateral epicondylitis; Tennis Elbow; Sustained stretch; Mobilization with Movement; Muscle strength
MeSH Terms: conditions — Tennis Elbow | interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The group will engage in traditional tennis elbow exercises and mobilization through movement.
  Interventions: Other: Mobilization with Movement
- Group B (Active Comparator): The group will be given a prolonged stretch along with conventional tennis elbow exercises.
  Interventions: Other: Sustained Stretch

INTERVENTIONS:
Other: Mobilization with Movement — Mobilization with Movement (MWM) is a manual therapy technique that combines active, patient-directed movements with passive joint mobilization to treat tennis elbow. To find joint restrictions or dysfunctions, a comprehensive patient assessment is the first step in the process. While the patient was in a supine position with the elbow fully extended and the forearm pronated, the therapist applied a sustained lateral glide of the forearm and stabilized the distal portion of the arm. While the patient asked to make a fist, the therapist kept up the lateral glide. Each session included three sets of movement-based mobilizations, each with ten repetitions. The entire course of treatment consists of twelve sessions.
  Arms: Group A
Other: Sustained Stretch — The basic concept of stretching involves lengthening the tendon during a state of relaxation. To stretch the Extensor Carpi Radialis Brevis tendon, the following position should be adopted: the elbow should be extended, the forearm in a pronated position, the wrist flexed, and the wrist should also be ulnar deviated, based on the patient's comfort level. This position should be maintained for 30 to 45 seconds and repeated three times before and after exercises in each treatment session, with a 30-second rest period in between.
  Arms: Group B

SUMMARY:
Tennis elbow, clinically known as lateral epicondylitis, is a prevalent musculoskeletal issue marked by pain and tenderness on the outer part of the elbow. It primarily affects the extensor tendon at the lateral epicondyle and is commonly linked to repetitive arm movements and overuse. Various treatment options are available for this condition, with two notable methods being sustained stretching and Mobilization with Movement (MWM). Sustained stretching involves holding the affected muscles and tendons in an extended position for a prolonged time to ease muscle tightness and enhance flexibility. Conversely, MWM integrates specific joint movements with the active involvement of the patient to improve joint mobility and reduce pain. Muscle strength plays a crucial role in the overall function of the upper limb, and enhancing this can positively affect daily activities. Furthermore, functional disability indicates how tennis elbow impacts a person's capacity to carry out everyday tasks.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at Riphah Rehab center over duration of eight months. The sample size will consist of 58 participants. Participants which meet the inclusion criteria will be taken through non-probability convenience sampling technique. 29 Participants will be assigned to Group A 29 to group B. Data will be collected using various assessment tools, including NPRS, ULFI, Universal Goniometer, Hand Held Dynamometer. Pre-intervention assessments will be conducted for groups. Data analysis will be performed by using SPSS 26 software.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females are affected. diagnosed with tennis elbow, characterized by pain and weakness on the outer side of the elbow.
* The pain has persisted for at least 4 to 6 months.
* Individuals experience difficulty gripping and lifting objects due to elbow pain.
* Positive results were observed in both the Mills and Cozen tests.

Exclusion Criteria:

* Presence of nerve injuries or neuropathies in the arm or hand.
* No history of recent trauma or fracture to the elbow.
* No neurological conditions affecting the arm or hand
* Acute inflammation or signs of infection in the elbow joint.
* Presence of cervical radiculopathy, thoracic outlet syndrome any systemic diseases

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pain: Numeric Pain Rating Scale (NPRS) | 4th week
  The most widely used pain rating scale, the Numeric Rating Scale (NPRS), has a range of 0 (no pain) to 10 (worst pain). The NPRS will be used to measure the degree of pain. For patients with tennis elbow, it will serve as an outcome measure. The NPRS is regarded as a valid, responsive, and dependable pain scale.
Function: Upper Limb Functional Index (ULFI) | 4th week
  Twenty-five items on the ULFI measure how patients with ULMSDs perceive their own limitations in their activities. Three possible answers are provided for each item: "Yes" (1 point), "Partly" (0.5 points), and "No" (0 points). The maximum disability is determined by multiplying the total points (ranging from 0 to 25) by 4. The patient's functional score in relation to their maximum or pre-injury function is then calculated by subtracting this total score from 100 (0% represents maximum limitation, 100% represents normal or pre-injury function). The total rating can be calculated with no more than two missing responses.
ROM: Universal Goniometer | 4th week
  A double-arm plastic goniometer with a semicircular scale is the most common goniometer for determining range of motion. We will measure the following wrist and elbow movements: wrist flexion, extension, radial and ulnar deviation, and elbow extension and pronation. Three measurements of each movement will be made, and the average will be computed for the outcome analysis.
Strength: Handheld Dynamometer: | 4th week
  A handheld dynamometer (CAMRY EH 101 Electronic Handheld Dynamometer) was used to measure grip strength. The American Society of Hand Therapists' measurement protocols were modified to place participants in a high sitting position, maintain an elbow at a slight 40° flexion, and adjust the handle to the second position. After thoroughly explaining the procedure, the patient was instructed to exert the greatest amount of force possible on the handle and maintain that position for three to five seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehab center., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karbowiak M, Holme T, Thambyrajah J, Di Mascio L. Management of lateral epicondylitis (tennis elbow). BMJ. 2023 May 18;381:e072574. doi: 10.1136/bmj-2022-072574. No abstract available. PMID 37201946
- [Background] Cutts S, Gangoo S, Modi N, Pasapula C. Tennis elbow: A clinical review article. J Orthop. 2019 Aug 10;17:203-207. doi: 10.1016/j.jor.2019.08.005. eCollection 2020 Jan-Feb. PMID 31889742
- [Background] Johns N, Shridhar V. Lateral epicondylitis: Current concepts. Aust J Gen Pract. 2020 Nov;49(11):707-709. doi: 10.31128/AJGP-07-20-5519. PMID 33123709
- [Background] Lenoir H, Mares O, Carlier Y. Management of lateral epicondylitis. Orthop Traumatol Surg Res. 2019 Dec;105(8S):S241-S246. doi: 10.1016/j.otsr.2019.09.004. Epub 2019 Sep 19. PMID 31543413
- [Background] Ma KL, Wang HQ. Management of Lateral Epicondylitis: A Narrative Literature Review. Pain Res Manag. 2020 May 5;2020:6965381. doi: 10.1155/2020/6965381. eCollection 2020. PMID 32454922
- [Background] Kjaer M. Role of extracellular matrix in adaptation of tendon and skeletal muscle to mechanical loading. Physiol Rev. 2004 Apr;84(2):649-98. doi: 10.1152/physrev.00031.2003. PMID 15044685
- [Background] Pathan AF, Sharath HV. A Review of Physiotherapy Techniques Used in the Treatment of Tennis Elbow. Cureus. 2023 Oct 26;15(10):e47706. doi: 10.7759/cureus.47706. eCollection 2023 Oct. PMID 38021828
- [Background] Reyhan AC, Sindel D, Dereli EE. The effects of Mulligan's mobilization with movement technique in patients with lateral epicondylitis. J Back Musculoskelet Rehabil. 2020;33(1):99-107. doi: 10.3233/BMR-181135. PMID 31104005
- [Background] Girgis B, Duarte JA. Efficacy of physical therapy interventions for chronic lateral elbow tendinopathy: a systematic review. Physical Therapy Reviews. 2020;25(1):42-59.